CLINICAL TRIAL: NCT04228718
Title: The Burden of Primary Caregivers of Spinal Muscular Atrophy Patients and Their Needs
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.728
Record Dates: First submitted 2020-01-12; First posted 2020-01-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-01

CONDITIONS: Spinal Muscular Atrophy; Caregiver Burden
Keywords: Spinal Muscular Atrophy; Caregiver Burden; Disabled persons; Caregivers
MeSH Terms: conditions — Muscular Atrophy, Spinal; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Zarit Burden Interview Scale — It is a questionnaire consisting of 22 items. A minimum score of 0 and a maximum score of 88 can be obtained. The higher the scale score, the higher the difficulty experienced.
Behavioral: Family Needs Survey (FNS) — It is a questionnaire consisting of 35 items prepared to determine the requirements. In the FNS survey; The points given to the items can be directly collected and the amount of family needs can be determined over the total score. The lowest score that can be obtained from FNS is 29 and the highest score is 87. As the scores obtained from the scale and subscales increase, it can be said that the families' level of necessity increases.
Other: Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) — CHOP-INTEND uses a scale of 0-64 points. Higher scores indicate better motor function. It is used to reliably measure natural motor function decline in infants with SMA Type 1.
Other: Hammersmith Functional Motor Scale Expanded (HMFSE) — It is an extended version of the 20-item HFMS. Based on another scale known as GMFM, 13 items were added and expanded HFMS to include these elements. Therefore, HFMSE is a scale used to evaluate motor functions in types 2 and 3 SMA. It contains 33 items with a total score of 66 on a scale of 0, 1, 2.

SUMMARY:
The purpose of this study is to assess carer burden, needs, and expectations of Spinal Muscular Atrophy Parents

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is a group of neuromuscular diseases involving the spinal cord anterior horn cells and brain stem motor nuclei. It is followed by programmed cell death. It progresses with symmetrical weakness and atrophy of voluntary muscles throughout the body. It leads to a decrease in mobility with progressive loss of power, and pulmonary function impairment with the involvement of the respiratory muscles.

Families who are confronted with these problems that arise after the birth of the baby or shortly after birth have a serious adaptation problem. When the course of the disease and its incurability are explained, patients and their families are under severe stress. Physical and emotional health is worse than normal healthy growing children's parents.

They need information, psychological and social support. The role of the family is very important in the life of children with disabilities. Family-oriented care; has been developed to facilitate the care process of children with special needs and to help their families. The main characteristics of the family-oriented approach are that families know their children in the best way, that each family is unique and different, and that family and community support is provided for the child's functionality. The assessment of family function helps the planning and management of treatment according to the concerns of the family. The education of the family, the socio-cultural structure and the psychological approach of the parents play an important role in the development of the child with SMA.

The aim of this study was to evaluate the care burden, needs and expectations of SMA parents and to reveal the problems clearly; so that this information can be used in rehabilitation planning and interpretation of results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with spinal muscular atrophy at between the ages of 0-18
2. Agree to participate in the study

Exclusion Criteria:

1-Refuse to participate in the study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with SMA type 1, type 2 or type 3 between the ages of 0-18 and their caregivers.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Zarit Burden Interview Scale | Day 0
  It is a questionnaire consisting of 22 items. A minimum score of 0 and a maximum score of 88 can be obtained. The higher the scale score, the higher the difficulty experienced.
Family Needs Survey (FNS) | Day 0
  It is a questionnaire consisting of 35 items prepared to determine the requirements. In the FNS survey; The points given to the items can be directly collected and the amount of family needs can be determined over the total score. The lowest score that can be obtained from FNS is 29 and the highest score is 87. As the scores obtained from the scale and subscales increase, it can be said that the families' level of necessity increases.

SECONDARY OUTCOMES:
Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) | Day 0
  CHOP-INTEND uses a scale of 0-64 points. Higher scores indicate better motor function. It is used to reliably measure natural motor function decline in infants with SMA Type 1.
Hammersmith Functional Motor Scale Expanded (HMFSE) | Day 0
  It is an extended version of the 20-item HFMS. Based on another scale known as Gross Motor Function Measure, 13 items were added and expanded HFMS to include these elements. Therefore, HFMSE is a scale used to evaluate motor functions in types 2 and 3 SMA. It contains 33 items with a total score of 66 on a scale of 0, 1, 2.

CONTACTS AND LOCATIONS:
Overall Officials: Naime Evrim Karadag Saygi, Prof, Study Director — Department of PM&R, Marmara University School of Medicine; Ayca Evkaya, Res. Asst., Principal Investigator — Department of Physiotherapy and Rehabilitation, Maltepe University
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Flunt D, Andreadis N, Menadue C, Welsh AW. Clinical commentary: obstetric and respiratory management of pregnancy with severe spinal muscular atrophy. Obstet Gynecol Int. 2009;2009:942301. doi: 10.1155/2009/942301. Epub 2009 May 19. PMID 19960049
- [Background] Pearn J. Incidence, prevalence, and gene frequency studies of chronic childhood spinal muscular atrophy. J Med Genet. 1978 Dec;15(6):409-13. doi: 10.1136/jmg.15.6.409. PMID 745211
- [Background] Strober JB, Tennekoon GI. Progressive spinal muscular atrophies. J Child Neurol. 1999 Nov;14(11):691-5. doi: 10.1177/088307389901401101. PMID 10593543
- [Background] Wirth B, Brichta L, Schrank B, Lochmuller H, Blick S, Baasner A, Heller R. Mildly affected patients with spinal muscular atrophy are partially protected by an increased SMN2 copy number. Hum Genet. 2006 May;119(4):422-8. doi: 10.1007/s00439-006-0156-7. Epub 2006 Mar 1. PMID 16508748
- [Background] Ho HM, Tseng YH, Hsin YM, Chou FH, Lin WT. Living with illness and self-transcendence: the lived experience of patients with spinal muscular atrophy. J Adv Nurs. 2016 Nov;72(11):2695-2705. doi: 10.1111/jan.13042. Epub 2016 Jun 30. PMID 27293032
- [Background] Finkel RS, McDermott MP, Kaufmann P, Darras BT, Chung WK, Sproule DM, Kang PB, Foley AR, Yang ML, Martens WB, Oskoui M, Glanzman AM, Flickinger J, Montes J, Dunaway S, O'Hagen J, Quigley J, Riley S, Benton M, Ryan PA, Montgomery M, Marra J, Gooch C, De Vivo DC. Observational study of spinal muscular atrophy type I and implications for clinical trials. Neurology. 2014 Aug 26;83(9):810-7. doi: 10.1212/WNL.0000000000000741. Epub 2014 Jul 30. PMID 25080519